CLINICAL TRIAL: NCT03931837
Title: Efficacy Testing of Different Tourniquet Pressure Used for Postoperative Pain Reduction in Total Knee Arthroplasty: A Prospective, Randomized Controlled Trials
Brief Title: Efficacy Testing of Different Tourniquet Pressure Used for Postoperative Pain Reduction in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Thammasat University (Other)
Collaborators: Boontanapibul, Krit, M.D. (Individual)
Responsible Party: Principal Investigator, piya pinsornsak, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTU-EC-OT-1-183/60
Record Dates: First submitted 2019-04-16; First posted 2019-04-30 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Tourniquet; Total knee arthroplasty; Postoperative pain; Range of motion; Wound complication
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tourniquet: Systolic blood pressure + 75 mmHg (Experimental): Before skin incision
  Interventions: Device: Tourniquet: Systolic blood pressure + 75 mmHg
- Tourniquet: Systolic blood pressure + 100 mmHg (Experimental): Before skin incision
  Interventions: Device: Tourniquet: Systolic blood pressure + 100 mmHg
- Tourniquet: Systolic blood pressure + 150 mmHg (Experimental): Before skin incision
  Interventions: Device: Tourniquet: Systolic blood pressure + 150 mmHg

INTERVENTIONS:
Device: Tourniquet: Systolic blood pressure + 75 mmHg — Spinal block without morphine. Medial parapatellar approach. Same posterior stabilized design and operated by a single surgeon. Drug: Peri-articular Transmine(15 mg/kg) combined with multimodal local anesthetic infiltration (0.5% bupivacaine 100 mg, morphine sulfate 5 mg, 0.1% epinephrine 0.6 mg, and ketorolac 30 mg) mixed NSS up to 75 mL. Procedure/Surgery: TXA combined with multimodal local anesthetic infiltration inject into peri-articular area (Anterior soft tissue 25 mL+Medial gutter area 25 mL+Lateral gutter area 25 mL) prior to capsular closure and tourniquet deflation
  Arms: Tourniquet: Systolic blood pressure + 75 mmHg
Device: Tourniquet: Systolic blood pressure + 100 mmHg — Spinal block without morphine. Medial parapatellar approach. Same posterior stabilized design and operated by a single surgeon. Drug: Peri-articular Transmine(15 mg/kg) combined with multimodal local anesthetic infiltration (0.5% bupivacaine 100 mg, morphine sulfate 5 mg, 0.1% epinephrine 0.6 mg, and ketorolac 30 mg) mixed NSS up to 75 mL. Procedure/Surgery: TXA combined with multimodal local anesthetic infiltration inject into peri-articular area (Anterior soft tissue 25 mL+Medial gutter area 25 mL+Lateral gutter area 25 mL) prior to capsular closure and tourniquet deflation
  Arms: Tourniquet: Systolic blood pressure + 100 mmHg
Device: Tourniquet: Systolic blood pressure + 150 mmHg — Spinal block without morphine. Medial parapatellar approach. Same posterior stabilized design and operated by a single surgeon. Drug: Peri-articular Transmine(15 mg/kg) combined with multimodal local anesthetic infiltration (0.5% bupivacaine 100 mg, morphine sulfate 5 mg, 0.1% epinephrine 0.6 mg, and ketorolac 30 mg) mixed NSS up to 75 mL. Procedure/Surgery: TXA combined with multimodal local anesthetic infiltration inject into peri-articular area (Anterior soft tissue 25 mL+Medial gutter area 25 mL+Lateral gutter area 25 mL) prior to capsular closure and tourniquet deflation
  Arms: Tourniquet: Systolic blood pressure + 150 mmHg

SUMMARY:
Tourniquet use during total knee replacement (TKR) improves visibility, significantly decreases intra-operative blood loss and reduce operative time. However, tourniquet use also has a negative effect on postoperative pain, postoperative range of motion(ROM), wound complication, deep vein thrombosis (DVT), pulmonary embolism (PE), thigh muscle strength, and functional recovery after TKR. Therefore, the investigators conducted a three-arm prospective, randomized, controlled trial study to compare the efficacy of different tourniquet pressure used between systolic blood pressure + 75 mmHg, systolic blood pressure + 100 mmHg, and systolic blood pressure + 150 mmHg.

DETAILED DESCRIPTION:
Patients scheduled for unilateral primary TKA; 150 patients were randomly assigned to receive tourniquet pressure used of systolic blood pressure + 75 mmHg, systolic blood pressure + 100 mmHg, and systolic blood pressure + 150 mmHg.

All patients had spinal anesthesia, the same operative procedure, and postoperative pain protocol. A visual analogue scale (VAS) for pain were recorded 24, 48 hours, and 2 weeks postoperatively. Quality of bloodless visual field and calculated blood loss were evaluated perioperatively. Postoperative ROM, wound complication, deep vein thrombosis (DVT), pulmonary embolism (PE) were recorded at 2, 6, and 12 weeks. Furthermore, Knee Society Score (KSS) also recorded at 6 weeks, 3 and 6 months. The reviewers were blinded to the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with osteoarthritis in need of a TKR

Exclusion Criteria:

* Inflammatory arthritis
* Post-traumatic arthritis
* Body mass index > 30 Kg/m2
* A history of or current venous thromboembolic disease
* Any underlying disease of hemostasis, cirrhosis, chronic renal failure, patients on anticoagulants or strong antiplatelet drugs (e.g. warfarin, clopidogrel)
* Preoperative hemoglobin <10 g/dL or a platelet count < 140,000 /uL3
* Allergy to transamine

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative visual analogue scale for pain | 48 hours after operation
  (VAS, 0 = no pain, 10 = the worst imaginable pain)

SECONDARY OUTCOMES:
Quality of bloodless visual field | Intraoperative evaluation
  (QBF, 0 = the worst quality, 10 = the best quality)
Changes from baseline hemoglobin concentrations | 48 hours after operation
Postoperative range of motion | 2 weeks, 6 weeks and 12 weeks
  Record with long arm goniometer
Number of patient with local soft tissue complications | 14 days after the operation
Number of patient with venous thromboembolism | 14 days after the operation
Knee society score | 6 weeks, 12 weeks and 6 months
  Score from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions

CONTACTS AND LOCATIONS:
Overall Officials: Piya Pinsornsak, Principal Investigator — Thammasat University Hospital
Locations (1):
- Thammasat university hospital, Pathum Thani, Klongluang, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi YJ, Ra HJ. Patient Satisfaction after Total Knee Arthroplasty. Knee Surg Relat Res. 2016 Mar;28(1):1-15. doi: 10.5792/ksrr.2016.28.1.1. Epub 2016 Feb 29. PMID 26955608
- [Background] Norton MR, Eyres KS. Irrigation and suction technique to ensure reliable cement penetration for total knee arthroplasty. J Arthroplasty. 2000 Jun;15(4):468-74. doi: 10.1054/arth.2000.2965. PMID 10884207
- [Background] Majkowski RS, Bannister GC, Miles AW. The effect of bleeding on the cement-bone interface. An experimental study. Clin Orthop Relat Res. 1994 Feb;(299):293-7. PMID 8119032
- [Background] Juliusson R, Arve J, Ryd L. Cementation pressure in arthroplasty. In vitro study of cement penetration into femoral heads. Acta Orthop Scand. 1994 Apr;65(2):131-4. doi: 10.3109/17453679408995419. PMID 8197842
- [Background] Walker PS, Soudry M, Ewald FC, McVickar H. Control of cement penetration in total knee arthroplasty. Clin Orthop Relat Res. 1984 May;(185):155-64. PMID 6705374
- [Background] Tetro AM, Rudan JF. The effects of a pneumatic tourniquet on blood loss in total knee arthroplasty. Can J Surg. 2001 Feb;44(1):33-8. PMID 11220796
- [Background] Ejaz A, Laursen AC, Kappel A, Laursen MB, Jakobsen T, Rasmussen S, Nielsen PT. Faster recovery without the use of a tourniquet in total knee arthroplasty. Acta Orthop. 2014 Aug;85(4):422-6. doi: 10.3109/17453674.2014.931197. Epub 2014 Jun 23. PMID 24954487
- [Background] Zhang W, Li N, Chen S, Tan Y, Al-Aidaros M, Chen L. The effects of a tourniquet used in total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2014 Mar 6;9(1):13. doi: 10.1186/1749-799X-9-13. PMID 24602486
- [Background] Lohmann-Jensen R, Holsgaard-Larsen A, Emmeluth C, Overgaard S, Jensen C. The efficacy of tourniquet assisted total knee arthroplasty on patient-reported and performance-based physical function: a randomized controlled trial protocol. BMC Musculoskelet Disord. 2014 Mar 29;15:110. doi: 10.1186/1471-2474-15-110. PMID 24678741
- [Background] Abdel-Salam A, Eyres KS. Effects of tourniquet during total knee arthroplasty. A prospective randomised study. J Bone Joint Surg Br. 1995 Mar;77(2):250-3. PMID 7706340
- [Background] Mori N, Kimura S, Onodera T, Iwasaki N, Nakagawa I, Masuda T. Use of a pneumatic tourniquet in total knee arthroplasty increases the risk of distal deep vein thrombosis: A prospective, randomized study. Knee. 2016 Oct;23(5):887-9. doi: 10.1016/j.knee.2016.02.007. Epub 2016 Jun 29. PMID 27372555
- [Background] Kumar N, Yadav C, Singh S, Kumar A, Vaithlingam A, Yadav S. Evaluation of pain in bilateral total knee replacement with and without tourniquet; a prospective randomized control trial. J Clin Orthop Trauma. 2015 Jun;6(2):85-8. doi: 10.1016/j.jcot.2015.01.095. Epub 2015 Feb 24. PMID 25983513
- [Background] Liu D, Graham D, Gillies K, Gillies RM. Effects of tourniquet use on quadriceps function and pain in total knee arthroplasty. Knee Surg Relat Res. 2014 Dec;26(4):207-13. doi: 10.5792/ksrr.2014.26.4.207. Epub 2014 Dec 2. PMID 25505702
- [Background] Torres PA, Helmstetter JA, Kaye AM, Kaye AD. Rhabdomyolysis: pathogenesis, diagnosis, and treatment. Ochsner J. 2015 Spring;15(1):58-69. PMID 25829882
- [Background] Sharma JP, Salhotra R. Tourniquets in orthopedic surgery. Indian J Orthop. 2012 Jul;46(4):377-83. doi: 10.4103/0019-5413.98824. PMID 22912509
- [Background] Ishii Y, Matsuda Y. Effect of tourniquet pressure on perioperative blood loss associated with cementless total knee arthroplasty: a prospective, randomized study. J Arthroplasty. 2005 Apr;20(3):325-30. doi: 10.1016/j.arth.2004.10.001. PMID 15809950
- [Background] Worland RL, Arredondo J, Angles F, Lopez-Jimenez F, Jessup DE. Thigh pain following tourniquet application in simultaneous bilateral total knee replacement arthroplasty. J Arthroplasty. 1997 Dec;12(8):848-52. doi: 10.1016/s0883-5403(97)90153-4. PMID 9458249